CLINICAL TRIAL: NCT04446013
Title: Comparison of Optic Nerve Sheath Diameter and Cerebral Regional Oxygen Saturation Measurements Between General and Spinal Anesthesia Applications in C-Section
Brief Title: Comparison of ONSD and rSO2 Measurements Between General and Spinal Anesthesia in C-Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020.05.1.16.048
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Intracranial Pressure Increase
Keywords: optic nerve sheath diameter; intracranial pressure; intraabdominal pressure; cerebral regional oxygen saturation; c-section
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group General Anesthesia (Experimental): C-Section under general anesthesia
  Interventions: Other: Optic Nerve Sheath Diameter Measurement
- Grup Spinal Anesthesia (Experimental): C-Section under spinal anesthesia
  Interventions: Other: Optic Nerve Sheath Diameter Measurement

INTERVENTIONS:
Other: Optic Nerve Sheath Diameter Measurement — The change in intracranial pressure via optic nerve sheath diameter measurement

SUMMARY:
General anesthesia and regional anesthesia can be chosen in cesarean operations. Endotracheal intubation and mechanical ventilation are components of general anesthesia. Endotracheal intubation has been shown to cause increased intracranial pressure. There is not enough information about the effect of spinal anesthesia on intracranial pressure during cesarean operations. Increased intracranial pressure can cause neurological complications by disrupting brain perfusion. For this reason, the investigators think that the safe anesthesia method should be determined especially in pregnant patients who are at risk of increased intracranial pressure.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective c-section operation
* Age between 18-49
* ASA I-II
* Gestational week ≥ 36

Exclusion Criteria:

* Ophthalmologic disease and optic nerve pathology
* Increased intracranial pressure
* History of cerebrovascular disease
* Cases where spinal anesthesia is contraindicated
* Emergency cesarean category level 1

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant and undergoing c-section operation
Enrollment: 81 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Optic Nerve Sheath Diameter | Throughout the surgery
  The change in intracranial pressure via optic nerve sheath diameter measurement during c-section among 5 time point.
Change in regional cerebral oxygen saturation | Throughout the surgery
  The change in regional cerebral oxygen saturation during c-section among 5 time point.

SECONDARY OUTCOMES:
Perioperative Hemodynamic Parameters | Throughout the surgery
  Mean arterial pressure in mmHg
Perioperative Hemodynamic Parameters | Throughout the surgery
  Heart rate beat per minute

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Can Tunalı, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Geeraerts T, Merceron S, Benhamou D, Vigue B, Duranteau J. Non-invasive assessment of intracranial pressure using ocular sonography in neurocritical care patients. Intensive Care Med. 2008 Nov;34(11):2062-7. doi: 10.1007/s00134-008-1149-x. Epub 2008 May 29. PMID 18509619
- [Background] Bauerle J, Nedelmann M. Sonographic assessment of the optic nerve sheath in idiopathic intracranial hypertension. J Neurol. 2011 Nov;258(11):2014-9. doi: 10.1007/s00415-011-6059-0. Epub 2011 Apr 28. PMID 21523461
- [Background] Yoshitani K, Kawaguchi M, Miura N, Okuno T, Kanoda T, Ohnishi Y, Kuro M. Effects of hemoglobin concentration, skull thickness, and the area of the cerebrospinal fluid layer on near-infrared spectroscopy measurements. Anesthesiology. 2007 Mar;106(3):458-62. doi: 10.1097/00000542-200703000-00009. PMID 17325503